CLINICAL TRIAL: NCT04728607
Title: Use of a Compression Device for Ring Removal: A Prospective Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1025977
Record Dates: First submitted 2020-10-14; First posted 2021-01-28 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Wounds and Injuries; Hand Injuries; Device Malfunction
MeSH Terms: conditions — Wounds and Injuries; Hand Injuries | interventions — Intermittent Pneumatic Compression Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants (Experimental): Individuals requiring ring removal.
  Interventions: Device: Compression device.

INTERVENTIONS:
Device: Compression device. — A compression device is a device that uses circumferential compression to reduce swelling around a stuck ring. The device is used by placing it near, but not overtop, the offending ring, and then is inflated compressing the finger. The device is applied, and the hand elevated, for approximately five minutes. The device is then removed, and with a small amount of lubricant, the ring is removed.

SUMMARY:
The usual treatment for stuck rings includes a variety of techniques including use of ice to reduce swelling, use of lubricants, and sometimes the use of string or ring cutters. The success rate of these techniques is variable and cutting the ring is usually reserved as a last resort. Sometimes removal of a ring can take time, and can cause some small injury to the patient. Because of this, it is important to consider other methods for ring removal.

This study is looking at using a device that uses compression to reduce swelling of the finger causing the ring to be stuck. This device has been approved for use in Canada. The purpose of this study is to evaluate how effective a compression device is at removing stuck rings.

The study question is: how effective is a compression device at removing stuck rings?

A Compression Device (CD) is a device that uses circumferential compression to reduce swelling around a stuck ring. The device is used by placing it near, but not over-top, the offending ring, and then is inflated compressing the finger. The device is applied, and the hand elevated, for approximately five minutes. The device is then removed, and with a small amount of lubricant, the ring is removed.

All patients requiring ring removal at the QEII emergency department, if a compression device can be used safely, will be asked if they would like to be included in the study and have their ring removal attempted by a compression device.

Following removal attempt, the clinician will document information about the ring removal. This will include some questions regarding the patient's experience with the removal. No identifying information or personal health information will be recorded.

The investigators plan to collect information about use of the compression device for a period of one year. Following this time, the data will be analyzed to determine how effective the compression device is at removing rings including statements regarding patient experience. This information will be documented in a manuscript intended for publication and may be presented at academic conferences or other continuing education events.

The investigators will be measuring the success rate of ring removal with the compression device.

In addition, the investigators will record information on any side effects of use of the compression device, as well as patient experience including pain and satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Individuals presenting to the QEII emergency department with a chief complaint of a stuck ring on a finger, or with heath conditions that necessitate removal of a ring that cannot be removed without clinician assistance.

Exclusion Criteria:

* Contraindications to compression device use including certain bone, nerve or blood vessel conditions.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-07-26 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Number of patients with successful ring removal using a compression device | 1 year
  Successful ring removal with compression device

CONTACTS AND LOCATIONS:
Locations (1):
- Dalhousie University, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No